CLINICAL TRIAL: NCT06366022
Title: Evaluation of the Treatment of Multiple Gingival Recession Using Modified Coronally Advanced Tunnel With Subepithelial Connective Tissue Graft Depending on the Positioning of the Graft
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Warsaw.06
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Gingival Recession
Keywords: tunneling technique
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multiple adjacent recessions coverage with sCTG with inner side of the graft (Experimental): Experimental: Multiple adjacent recessions coverage with subepithelial connective tissue graft..
  A modified microsurgical tunnel technique. Initial sulcular incisions with a microsurgical blade are followed by a full-thickness buccal flap preparations till muco-gingival junction using the tunneling knives. Subsequently, the split-thickness preparation is extended into the mucosal tissue to gain sufficient flap mobility. The papillary regions are detached in their buccal aspects with the periosteum. The graft is inserted the inner side into the tunnel and stabilized with absorbable suspensory sutures. The buccal flap is advanced coronally and stabilized with non-absorbable suspensory sutures.
  Interventions: Device: The tunnel technique for root coverage with CTG with inner side of the graft
- Multiple adjacent recessions coverage with sCTG with outer side of the graft (Active Comparator): Multiple adjacent recessions coverage with subepithelial connective tissue graft..
  A modified microsurgical tunnel technique. Initial sulcular incisions with a microsurgical blade are followed by a full-thickness buccal flap preparations till muco-gingival junction using the tunneling knives. Subsequently, the split-thickness preparation is extended into the mucosal tissue to gain sufficient flap mobility. The papillary regions are detached in their buccal aspects with the periosteum. The graft is inserted the outer side into the tunnel and stabilized with absorbable suspensory sutures. The buccal flap is advanced coronally and stabilized with non-absorbable suspensory sutures.
  Interventions: Device: The tunnel technique for root coverage with CTG with outer side of the graft

INTERVENTIONS:
Device: The tunnel technique for root coverage with CTG with inner side of the graft — Procedure: The tunnel technique for root coverage with CTG with inner side of the graft
  Arms: Multiple adjacent recessions coverage with sCTG with inner side of the graft
Device: The tunnel technique for root coverage with CTG with outer side of the graft — The tunnel technique for root coverage with CTG with outer side of the graft
  Arms: Multiple adjacent recessions coverage with sCTG with outer side of the graft

SUMMARY:
Microsurgical coronally advanced tunnel procedures using subepithelial connective tissue grafts (sCTG) are predictable for healing of multiple adjacent type 1 and 2 gingival recessions (RT1 and RT2). In order to reduce patient morbidity and enhance periodontal wound healing with sCTG can be used. The aim of this study is to compare the results of the modified tunneling technique with subepithelial connective tissue graft in gingival recessions placed with the inner side towards the flap cover graft and the outer side towards the flap cover graft.

DETAILED DESCRIPTION:
Condition or disease:Multiple Gingival Recession

Intervention/treatment:

Device: Modified coronally advanced tunnel with connective tissue graft placed with inner side towards the flap Device: Modified coronally advanced tunnel with subepithelial connective tissue graft with the outer side towards the flap Phase :Not Applicable

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Bilateral multiple gingival recessions in homologous teeth in the same arch.

Exclusion Criteria:

* Full-mouth plaque index ≥ 20% (Ainamo & Bay 1975)
* Full-mouth sulcus bleeding index ≥ 15% (Mühlemann & Son 1971)
* Smoking
* Systemic diseases with compromised healing potential of infectious diseases
* Drugs affecting periodontal health / healing
* Pregnant and lactating females
* Previous periodontal surgery in the area

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Clinical attachment level (CAL) | Time Frame: 6 months after surgery
  Distance from the cementoenamel junction to the bottom of the gingival sulcus
Recession height (RH) | Time Frame: 6 months after surgery
  Distance from the cementoenamel junction to the gingival margin
Recession width (RW) | Time Frame: 6 months after surgery
  Distance measured horizontally at cementoenamel junction level from one border of the recession to another
Width of keratinized tissue (KTW) | Time Frame: 6 months after surgery
  Distance between the most apical point of the gingival margin and the mucogingival junction
Thickness of keratinized tissue (GT | Time Frame: 6 months after surgery
  Thickness of the gingiva measured 2 mm apical to the gingival margin
Average recession coverage (ARC) | Time Frame: 6 months after surgery
  The percentage of covered recession area
Complete recession coverage | Time Frame: 6 months after surgery
  The percentage of sites with complete root coverage

SECONDARY OUTCOMES:
Probing pocket depth (PPD) | Time Frame: 6 months after surgery
  Distance from the gingival margin to the bottom of the gingival sulcus
Root coverage esthetic score (RES) | Time Frame: 6 months after surgery
  A score including root coverage, marginal gingival tissue contour, mucogingival junction alignment, soft tissue texture and gingival colour according to Cairo et al. (1999)
Post surgical pain and swelling | Time Frame:, 7 and 14 days after surgery
  Questionnaire about post surgical pain and swelling using a Visual Analog Scale with values 0 (no pain / swelling), 1, 2, 3, 4, 5(moderate pain/swelling), 6, 7, 8, 9, 10 (worst pain / swelling). Lower values represent lower post surgical discomfort and are considered better.
Patient's satisfaction with treatment | Time Frame: 6 months after surgery ]
  Questionnaire about patient's esthetic perception of gingiva and overall satisfaction using a Visual Analog Scale from 0 (dissatisfaction with esthetic outcome), 2, 3, 4, 5 (moderate satisfaction with easthetic outcome), 6, 7, 8, 9, 10 (best satisfaction with esthetic outcome). Higher values are considered better.

CONTACTS AND LOCATIONS:
Overall Officials: Bartłomiej Górski, PhD, Principal Investigator — Department of Periodontology and Oral Mucosa Diseases, Medical University of Warsaw
Locations (1):
- Department of Periodontology and Oral Mucosa Diseases, Medical University of Warsaw, Warsaw, MAzowsze, Poland